CLINICAL TRIAL: NCT03271762
Title: Multicentre and Randomized Study of MITRACLIP® Transcatheter Mitral Valve Repair in Patients With Severe Primary Mitral Regurgitation Eligible for High-risk Surgery
Brief Title: Multicentre Study of MITRACLIP® Transcatheter Mitral Valve Repair in Patients With Severe Primary Mitral Regurgitation Eligible for High-risk Surgery
Acronym: MITRA-HR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Ministère de la Santé (Unknown); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC17_0002
Record Dates: First submitted 2017-08-25; First posted 2017-09-05 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Mitral Regurgitation
Keywords: MITRACLIP; primary Mitral Regurgitation; high surgical risks
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MITRACLIP NT, MITRACLIP NTR/XTR, MITRACLIP G4NT/XT, MITRACLIP G4NTW/XTW Device (Experimental): MitraClip NT System includes a MitraClip device, a steerable guide catheter and a MitraClip delivery system
  Interventions: Device: percutaneous mitral valve repair with MITRACLIP NT, MITRACLIP NTR/XTR, MITRACLIP G4NT/XT, MITRACLIP G4NTW/XTW
- cardiac surgery (Active Comparator): mitral valve repair in first intervention, valve replacement if repair not feasible
  Interventions: Procedure: cardiac surgery

INTERVENTIONS:
Device: percutaneous mitral valve repair with MITRACLIP NT, MITRACLIP NTR/XTR, MITRACLIP G4NT/XT, MITRACLIP G4NTW/XTW — percutaneous mitral valve repair Percutaneous MitraClip Device Implantation
  Other Names: MITRACLIP
  Arms: MITRACLIP NT, MITRACLIP NTR/XTR, MITRACLIP G4NT/XT, MITRACLIP G4NTW/XTW Device
Procedure: cardiac surgery — mitral valve repair or mitral valve remplacement
  Arms: cardiac surgery

SUMMARY:
The objective of the study is to demonstrate the non-inferiority for clinical efficacy of an endovascular treatment strategy with the MitraClip® in comparison with a surgical treatment strategy in patients with severe primary mitral regurgitation judged eligible for anatomical repair with the MitraClip® or mitral valve surgery with high surgical risk.

This trial is a French and Monegasque, multicenter and randomized trial. Patients enrolled will be clinically followed for 2 years ( clinical visit at 1 month, at 6 months and 12 months, phone call at 18 months and clincial visit at 24 months).

ELIGIBILITY:
Inclusion Criteria:

Primary Mitral Regurgitation grade 3+ or 4+

* Patients in class II to IV NYHA
* Mitral valve anatomy appropriate to MitraClip® therapy and mitral valve surgery
* Adult patients judged eligible for mitral valve surgery by the local heart team but at high surgical risk defined as: age ≥ 75 years and STS score ≥ 6 % or one frailty index or one major organ system compromise or one possible procedure-specific impediment (using MVARC definitions) ; or age < 75 years and STS score > 8 % or at least one other high-risk criterion following the MVARC definitions; or age > 80 years and judged at high risk for surgery by the local heart team
* Isolated Mitral valve pathology
* If revascularization procedures are required, they must be performed more than 30 days from intervention (D0)
* Patients affiliate to social security

Non-inclusion Criteria:

* Life expectancy < 1 year due to non-cardiac conditions
* Secondary Mitral regurgitation
* Evolving endocarditis or active endocarditis or inflammatory disease in the last 3 months
* Patient who cannot tolerate procedural anticoagulation or post procedural antiplatelet regimen
* Rheumatic mitral valve disease
* Evidence of intracardiac, inferior vena cava or femoral venous thrombus
* Valve anatomy not compatible with MitraClip® implantation (cf. colum 3 table 3 page 57)
* Stroke or transient ischaemic event within 30 days before D0
* Modified Rankin Scale ≥4 disability (appendix 9)
* TAVR within 30 days before D0-Untreated, clinically significant coronary artery disease requiring revascularization
* Any percutaneous cardiovascular intervention within 30 days before D0 including ATC
* Cardiovascular surgery, or carotid surgery within 30 days before D0
* Any prior mitral valve surgery or transcatheter mitral valve procedure
* Need for any concomitant cardiac surgery including treatment of severe secondary tricuspid regurgitation in accordance with class I recommendation in 2017 ESC guidelines. Surgical treatment of mild or moderate secondary tricuspid regurgitation (Class IIa and IIb recommendations) can still be performed in the protocol according to the local heart team decison
* NYHA functional class I
* LVEF < 30%
* Primary MR grade 1 to 2
* Subjects in whom transesophageal echocardiography or transseptal catheterization are contraindicated or high-risk
* Any condition preventing the patient from completing all protocol procedures (including compliance with guidelines directed medical therapy) and follow-up visits
* Patient unable or unwilling to provide written, informed consent before study enrolment
* Pregnant or nursing women
* Vulnerable people: persons deprived of liberty; under trusteeship or under curatorship
* Participation in another trial that would interfere with this trial

Exclusion criteria

* Not eligible for a MitraClip® intervention after Core Lab evaluation
* Before randomization (D-21) the patient no longer fulfills eligibility criteria (inclusion criteria and non-inclusion criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2018-03-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality, unplanned hospitalizations for heart failure and mitral valve reintervention | 12 months
  comparison between arms of:
  * number and reason of death
  * number and reason unplanned rehospitalisation for cardiovascular reasons,
  * number of mitral valve reintervention

SECONDARY OUTCOMES:
occurrence of a major adverse event | 30 days
  all-cause death, need for non-elective cardiovascular or thoracic surgery, device or procedure-related adverse events, major bleeding complications or serious bleeding, major access site vascular complications, major cardiac structural complications, pulmonary complications (device or procedure-related), stroke and other cerebrovascular events, myocardial infarction, acute kidney injury or progression of chronic kidney disease, arrhythmias and conduction system disturbances, unplanned mitral valve surgery due to device/procedure failure or malfunction, requirement for valve replacement after valve repair failure, unplanned cardiac surgery for any cause

OTHER OUTCOMES:
Overall rate of surgery related Serious Adverse Events (SAEs) and Serious Adverse Device Effects (SADEs) Effects (SADEs) | 6, 12 and 24 months
  SAEs et SADEs rate related to protocol procedure all SAEs and SADEs
all-cause mortality | 30 days and 6, 12 and 24 months
  Rate of global mortality (all-causes)
cardiovascular mortality | 30 days and 6, 12 and 24 months
  Rate of cardiovascular mortality
unplanned heart failure rehospitalization | 6, 12 and 24 months
  Rate of unplanned heart failure rehospitalization
unplanned rehospitalization rate for cardiovascular reasons | 30 days 6, 12 and 24 months
  Rate of unplanned rehospitalization for cardiovascular reasons
mitral valve reintervention | 30 days 6, 12 and 24 months
  Mitral valve reintervention rate
residual MR | 30 days 6, 12 and 24 months
  MR (Mitral Regurgitation): grade
left and right chamber remodelling and parameters (dimension) | baseline, 30 days and 12 months
  End-systolic dimension End-diastolic dimension Left atrial dimension
left and right chamber remodelling and parameters (volume) | baseline, 30 days and 12 months
  End-systolic volume End-diastolic volume Left atrial volume
left ventricular ejection fraction modification | baseline, 30 days and 12 months
  Left ventricular ejection fraction
mitral valve remodelling | baseline, 30 days and 12 months
  Mitral valve area and mean gradient
Left atrial and pulmonary artery pressures | baseline, 30 days and 12 months
  Left atrial and pulmonary artery pressures
change in 6-minute Walking Test (functional evaluation) | baseline, 6 and 12 months
  6-minute Walking Test
surveillance of cardiac and renal function | baseline, 30 days, 6, 12 and 24 months
  NT ProBNP or BNP creatininemia, ureamia
change in Quality of Life scores | baseline, 30 days, 6, 12 and 24 months
  Quality of Life EQ-5D score SF-36 score
Cost-effectiveness analysis (economic efficiency) | 24 months
  Incremental cost-effectiveness ratio (cost per Quality-Adjusted Life-Year, QALY)

CONTACTS AND LOCATIONS:
Locations (31):
- France (31):
  - Chu Angers, Angers
  - Ch Annecy, Annecy
  - Chu Bordeaux, Bordeaux
  - Chru Brest, Brest
  - Hopital Henri Mondor Aphp, Créteil
  - Chu Grenoble, Grenoble
  - Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - Chru Lille, Lille
  - Hopital Prive Le Bois Lille, Lille
  - Clinique de La Sauvegarde, Lyon
  - CHU LYON, Lyon
  - Hopital La Timone, Marseille
  - Hopital St Joseph, Marseille
  - Institut Hospitalier Jacques Cartier, Massy
  - Clinique Du Millenaire, Montpellier
  - Chu Nantes, Nantes
  - Hopital Bichat, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital La Pitie Salpetriere, Paris
  - Institut Mutualiste Montsouris, Paris
  - Chu Poitiers, Poitiers
  - Chu Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU Félix Guyon, Saint-Denis
  - Centre Cardiologique Du Nord, Saint-Denis
  - Chu Saint Etienne, Saint-Etienne
  - Hopital Civil Strasbourg, Strasbourg
  - Clinique Pasteur, Toulouse
  - Hopital Rangueil, Toulouse
  - Chru Tours, Tours
  - Clinique Du Tonkin, Villeurbanne